CLINICAL TRIAL: NCT02752854
Title: Pain Threshold Measurements in High and Low Altitude Among Healthy Volunteer Adults: A Comparative Study
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Taif University (Other)
Responsible Party: Principal Investigator, Dr. Nashwa Sayed Hamed, Associate professor of physical therapy, Taif University
Other Study IDs: TU217; U1111-1181-8637 (Other: Universal Trial Number)
Record Dates: First submitted 2016-04-13; First posted 2016-04-27 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-04

CONDITIONS: Pain
Keywords: pain scores; pressure algometer; healthy volunteer adults
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group A: Pain threshold measurement in high altitude
  Interventions: Other: pain threshold measurement
- Group B: Pain threshold measurement in low altitude
  Interventions: Other: pain threshold measurement

INTERVENTIONS:
Other: pain threshold measurement — pressure algometer

SUMMARY:
one measurement of pain threshold in high altitude and in low altitude using pressure algometer and Situational pain scale.

DETAILED DESCRIPTION:
the aim of the study is to compare between pain threshold in high 1.9000 m above sea level and low altitude at sea level in healthy volunteer adults.

Assessment performed using:

1. pressure algometer.
2. situational pain scale

ELIGIBILITY:
Inclusion Criteria:

* age 18-52 years old.
* healthy volunteers

Exclusion Criteria:

* no musculoskeletal problems including muscle spasm
* no recent injuries or operations.
* not suffering from any painful condition.
* not on pain medications or antidepressant

Ages: 18 Years to 52 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: healthy volunteer adults
Sampling Method: Non-Probability Sample
Enrollment: 484 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-05 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Pain threshold assessed with a pressure algometer | 1 year
  pain threshold measurement

SECONDARY OUTCOMES:
situational pain scale | 1 year
  measures pain perception in different painful situations

CONTACTS AND LOCATIONS:
Overall Officials: Amro A Almaz, PhD, Study Chair — Head of scientific research board

IPD SHARING:
Plan to Share IPD: No